CLINICAL TRIAL: NCT00839345
Title: Resistance to Antiplatelet Agents, Its Etiology and the Possibility of Its Affection
Brief Title: Clopidogrel Resistance and the Possibility of Its Affection
Status: Temporarily not available | Type: Expanded Access
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, Associate professor, Charles University, Czech Republic
Other Study IDs: CLO-OSM-01
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: platelet; clopidogrel; VerifyNow; ticlopidine; thrombosis
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Clopidogrel

INTERVENTIONS:
Drug: clopidogrel — The intervention will involve the change of dosage or change of drug. The traditional maintenance dose of clopidogrel is 75 mg per day. We will test in non-responders to this classical dose higher doses up to 225mg per day. In patients,who will not respond to this 3times higher dose,clopidogrel will be replaced by ticlopidine.
  Other Names: Plavix

SUMMARY:
The purpose of the study is to determine, whether the resistance to clopidogrel could be affected by higher doses of this drug, or by replacement of clopidogrel with another ADP-antagonist ticlopidine.

DETAILED DESCRIPTION:
Patients after percutaneous coronary intervention (PCI) with stent implantation have to be treated by dual antiplatelet therapy, which standard part represents clopidogrel. The response to clopidogrel in population exhibits wide interindividual variability. According to some recent works, patients with clopidogrel resistance are in higher risk for recurrence of myocardial infarction in comparison with the patients with sufficient clopidogrel effectiveness. The treatment of clopidogrel resistance is still unknown. Our project should contribute to the better understanding of the clinical impact of clopidogrel resistance and its genetical determination. We will test the hypothesis, whether the clopidogrel resistance could be influenced by higher dose of this drug or by replacement to ticlopidine (ADP antagonist with different biotransformation in the liver). Therefore, 500 pts. will be tested to clopidogrel resistance. We expect 5-10% of resistent pts. This pts. will be treated by higher dose (150mg or 225mg/day) with repeated tests of clopidogrel effectiveness after each dose enhancement. If 225mg/day will be insufficient, clopidogrel will be replaced by ticlopidine with repeated test. We expect, that better definition of clinical and and genetic correlate of clopidogrel resistance will improve our knowledge of this disorder. Nevertheless, the achievement of sufficient effect of clopidogrel in some still resistant patients will lead to the improvement of the treatment

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* coronary artery disease verified by coronary angiography
* percutaneous coronary intervention with stent implantation
* standard indication for dual antiplatelet therapy

Exclusion Criteria:

* scheduled surgical revascularization by aortocoronary bypass
* insufficient cooperation of the patient
* coagulopathy in history with a higher risk of bleeding
* life expectancy shorter than 1 year
* severe anemia with hemoglobin level< 10,0 g/dl
* platelet count < 100,000)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, Dept. Of Cardiology, Charles University Hospital, Prague, Czechia